CLINICAL TRIAL: NCT07237503
Title: THE EFFECT OF CALISTHENIC EXERCISES ON FATIGUE AND EXERCISE ATTITUDES IN PATIENTS WITH LUNG CANCER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Kardelen HATIMOĞULLARI, specialist physiotherapist, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/051
Record Dates: First submitted 2025-07-07; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer (NSCLC); Physiotherapy; Fatigue in Cancer Survivors; Exercise
Keywords: Lung cancer, exercise, fatigue, physiotherapist
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Motor Activity; Fatigue | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: During the 8-week period, both groups completed exercise training three times a week at low to moderate intensity (50-60% of maximal heart rate). In the first week, patients in both groups were allowed to exercise as much as they could tolerate, with more frequent rest intervals provided. Starting from the third week, as patients' tolerance improved, rest intervals were reduced and the number of repetitions was adjusted to 10. By the second month, for patients who were able to tolerate more, the number of repetitions was increased to 12, and in the following week, exercises were planned as 2 sets for suitable patients.
  In the Physiotherapist-Led Exercise group, the exercise sessions were conducted under the supervision of a physiotherapist, and patients' respiratory rate, fatigue severity, blood pressure, and pain were regularly monitored.
  In the Home Exercise Training group, the same exercises were demonstrated practically during the first session, and patients were instructed to re
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapist-Led Exercise (Experimental): Patients in Group 1 were exercised 3 days a week for 8 weeks at 50-60% of maximal heart rate for 40 min, accompanied by a physiotherapist.
  Interventions: Behavioral: Exercise
- Home Exercise Group (Active Comparator): . Patients in Group 2 were given an exercise booklet and followed up with weekly controls.
  Interventions: Behavioral: Home based exercise

INTERVENTIONS:
Behavioral: Exercise — Patients in Group 1 were exercised 3 days a week for 8 weeks at 50-60% of maximal heart rate for 40 min, accompanied by a physiotherapist.
  Arms: Physiotherapist-Led Exercise
Behavioral: Home based exercise — Patients in Group 2 were given an exercise booklet and followed up with weekly controls.
  Arms: Home Exercise Group

SUMMARY:
Purpose: This study was carried out to investigate fatigue and exercise barriers of calisthenic exercises in patients with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-65
* Patients with lung cancer who continue to receive chemotherapy, radiotherapy or immunotherapy (smart drugs)
* Patients reporting fatigue of 3 or more on the Modified Borg Scale

Exclusion Criteria:

* Uncontrolled hypertension, diabetes mellitus, heart failure and atrial fibrillation
* Any acute infection at the time of assessment
* Those with orthopaedic, neurological, psychological, etc. problems that may limit the assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Exercise benefits and barriers | 2 month
  the perception of disability decreases in the group exercising with a physiotherapist

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu Üniversitesi, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No